CLINICAL TRIAL: NCT02061254
Title: Transient Elastography DEdicated to Cosmetology And Dermatology (TEDECAD)
Acronym: TEDECAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Echosens (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PFUI 2013 - AM / TEDECAD
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2015-08

CONDITIONS: Venous Insufficiency; Lymphedema
Keywords: Venous insufficiency; Lymphedema; Elastograph; Ultrasonography; Fibrosis; Dermis; Hypodermis; Skin
MeSH Terms: conditions — Venous Insufficiency; Lymphedema; Fibrosis | interventions — Ultrasonography; Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 groups of subjects (Experimental): 3 groups:
  * group of 48 healthy volunteers (matched with venous insufficiency patients)
  * group of 48 patients with venous insufficiency (16 with stage 1/2, 16 with stage 3/4, 16 with stage 5/6)
  * group of 40 patients with unilateral lymphedema (20 on upper limb (10 early stage, 10 severe stage), and 20 on lower limb (10 early stage, 10 severe stage))
  Each group have the same interventions: physical examination, measures by cutometer, high resolution ultrasonography, elastography 30 persons will have a skin biopsy (15 healthy volunteers and 15 patients with venous insufficiency) For patients with lymphedema, all measures will be performed on lymphedema limb and on controlateral healthy limb
  Interventions: Device: Cutometer; Device: High resolution ultrasonography (echography); Device: Elastography; Procedure: Skin biopsy

INTERVENTIONS:
Device: Cutometer — 3 measures by cutometer on each area: the mean value will be the final value
  Other Names: Cutometer MPA 580 (Monaderm)
Device: High resolution ultrasonography (echography) — Cutaneous echography on the 3 areas, in order to measure skin thickness and echogenicity Measures are blinded to cutometer (by a different investigator)
  Other Names: Dermcup (Atys medical)
Device: Elastography — 10 measures on the 3 areas (central measures will be doubled) Measures will be performed blinded to cutometer
  Other Names: high resolution elastography pulse
Procedure: Skin biopsy — Skin biopsy of 3 mm in diameter, for 30 participants, to evaluate histological fibrosis

SUMMARY:
Explorative study on a medical device with two steps. The first pilot step will be on 8 patients (4 with lymphedema and 4 with venous insufficiency). The main objective is to assess the feasibility of measures by high resolution transient elastography on these pathologic skins, and to define 3 areas for measures.

The second step will be on 136 participants (48 healthy volunteers, 48 with venous insufficiency and 40 with unilateral lymphedema of a limb). The main objective is to quantify, by high resolution transient elastography, the dermal and hypodermal cutaneous fibrosis in limbs with lymphedema and venous insufficiency, and to compare it to healthy skin.

DETAILED DESCRIPTION:
This diagnostic study will be performed in two steps, in the goal of evaluating a new device, called elastograph.

The first pilot step will be on 8 patients (4 with lymphedema and 4 with venous insufficiency). The main objective is to assess the feasibility of measures by high resolution transient elastography on these pathologic skins, and to define 3 areas for measures.

The second step will be on 136 participants (48 healthy volunteers, 48 with venous insufficiency and 40 with unilateral lymphedema of a limb). The main objective is to quantify, by high resolution transient elastography, the dermal and hypodermal cutaneous fibrosis in limbs with lymphedema and venous insufficiency, and to compare it to healthy skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients group

  * More than 18 years old
  * Inform consent form signed
  * Affiliated to medical insurance
  * No allergy to local anaesthetic drugs known
  * For patients with lymphedema of upper limb: unilateral lymphedema occurred after a surgery and/or radiotherapy clinically confirmed by a dermatologist or a physician trained to lymphology, or primitive lymphoedema clinically confirmed by a dermatologist or a physician trained to lymphology, whom the unilateral characteristic will be proved by a recent lymphoscintigraphy (less than 2 years)
  * For patients with lymphedema of lower limb: unilateral lymphedema occurred after a surgery and/or radiotherapy clinically confirmed by a dermatologist or a physician trained to lymphology, or primitive lymphoedema clinically confirmed by a dermatologist, whom the unilateral characteristic will be proved by a recent lymphoscintigraphy (less than 2 years)
  * For patients with venous insufficiency without leg ulcer: venous insufficiency without ulcer, clinically diagnosed by a dermatologist or a physician trained to angiology
  * For patients with venous insufficiency with ulcer: venous insufficiency with ulcer, clinically diagnosed by a dermatologist or a physician trained to angiology
* Healthy group

  * Healthy volunteer
  * More than 18 years-old
  * Without any cutaneous pathology on the studied areas
  * No venous insufficiency ; this will be confirmed by a physician trained to stages of venous insufficiency and will be defined by absence of: edema, varicosities, dilated veins, telangiectasia, venous dermatitis, sclerosis, leg ulcer
  * Inform consent form signed
  * Affiliated to medical insurance
  * No allergy to local anaesthetic drugs known
  * Matched according to age (± 10 years), gender and weight (± 20 kg) to patients with venous insufficiency

Exclusion Criteria:

* Patients group

  * History of aesthetic surgery on studied areas
  * Cutaneous abnormalities (including scars) on studied areas, except for signs of lymphedema or venous insufficiency
  * Acute or offset chronic pathology which doesn't allow long-timed explorations (according to investigator's assessment)
  * Inability to understand information and to sign the consent form (linguistics reasons or neuro-psychological)
  * Pregnant women, lactating women, and women in age for procreation and without reliable contraception or without history of hysterectomy
  * Person under guardianship
* Healthy group

  * Haemophilia or equivalent pathology
  * Cutaneous abnormalities on studied areas (including scars)
  * History of aesthetic surgery on studied areas
  * Acute or offset chronic pathology which doesn't allow long-timed explorations (according to investigator's assessment)
  * Inability to understand information and to sign the consent form (linguistics reasons or neuro-psychological)
  * Pregnant women, lactating women, and women in age for procreation and without reliable contraception or without antecedent of hysterectomy
  * Person under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assessment of dermal/hypodermal fibrosis in lymphedema and venous insuffisency | One day
  * Step 1: follow-up of the shear waves spreading, in cutaneous tissues, within 2-3 mm
  * Step 2: measure of fibrosis of the cutaneous tissue, by transient elastography (elastograph, in kPa)

SECONDARY OUTCOMES:
Cutaneous fibrosis measured by cutometer | One day
  Cutaneous fibrosis measured by cutometer
Cutaneous fibrosis assessed by histology | 12 months
  Cutaneous fibrosis assessed by histology (skin biopsies), using a semi-quantitative scale (0 to 3, from no fibrosis to major fibrosis) Analysis of the samples will be performed altogether at the end of inclusions.
Cutaneous thickness measured by high resolution ultrasonography | One day
  Cutaneous thickness measured by high resolution ultrasonography (in mm)
Clinical score of fibrosis | One day
  Clinical score of fibrosis, assessed by a scale from 0 (normal skin) to 3 (severe fibrosis): this score is derived from modified Rodnan skin score used in scleroderma
Echogenicity of the dermis and superficial hypodermis | One day
  Echogenicity of the dermis and superficial hypodermis assessed by high resolution ultrasonography
Assessement of adverse events | 15 days
  Assessement of adverse events (pain with a visual analogic scale from 0 to 100, infections of the site of skin biopsies, others)

CONTACTS AND LOCATIONS:
Overall Officials: Annabel MARUANI, MD, PhD, Principal Investigator — CHRU TOURS
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Result] Mofid Y, Faleweei G, Chartier C, Machet L, Vierron E, Gissot V, Tauveront V, Georgescou G, Dujardin PA, Machet MC, Kervarrec T, Patat F, Ossant F, Maruani A. High-Frequency Transient Elastography Prototype to Assess Skin (Dermis) Fibrosis: A Diagnostic Study in Patients with Venous Insufficiency and Controls. Ultraschall Med. 2021 Oct;42(5):503-513. doi: 10.1055/a-1047-3146. Epub 2020 Mar 18. PMID 32187631
- See also: Clinical Investigation Center - Technological Innovations — http://cic-it-tours.fr/